CLINICAL TRIAL: NCT00678301
Title: Primary Vaccination Course in Children Receiving the Pneumococcal Vaccine GSK 1024850A Co-administered With Zilbrix™ Hib and Polio Sabin™
Brief Title: Primary Vaccination Course in Children Receiving the Pneumococcal Vaccine GSK 1024850A, Zilbrix™ Hib and Polio Sabin™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110521; 2011-004650-25 (EudraCT Number)
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Infections, Streptococcal
Keywords: pneumococcal conjugate vaccine; Streptococcus pneumoniae
MeSH Terms: conditions — Streptococcal Infections

ARMS (2):
- SYNFLORIX™ + ZILBRIX™ HIB + POLIO SABIN™ (Experimental): Subjects in this group received 3 doses of Synflorix™ vaccine, according to a 3-dose schedule at 6-10-14 weeks of age co-administered with 3 doses of Expanded Program on Immunization (EPI) vaccines Zilbrix™ Hib and Polio Sabin™ according to the same schedule. The Synflorix™ and Zilbrix™ Hib vaccines were administered by intramuscular injection, in the right and left thigh respectively. The Polio Sabin™ vaccine was administered orally.
  Interventions: Biological: GSK Biologicals' Synflorix™; Biological: GSK Biologicals' Polio Sabin™; Biological: GSK Biologicals' Zilbrix™ Hib
- ZILBRIX™ HIB + POLIO SABIN™ (Experimental): Subjects in this group received 3 doses of Expanded Program on Immunization (EPI) vaccines Zilbrix™ Hib and Polio Sabin™ according to a 3-dose schedule at 6-10-14 weeks of age. The Zilbrix™ Hib vaccine was administered by intramuscular injection, in the left thigh. The Polio Sabin™ vaccine was administered orally.
  Interventions: Biological: GSK Biologicals' Polio Sabin™; Biological: GSK Biologicals' Zilbrix™ Hib

INTERVENTIONS:
Biological: GSK Biologicals' Synflorix™ — 3 IM doses.
  Other Names: 10Pn
  Arms: SYNFLORIX™ + ZILBRIX™ HIB + POLIO SABIN™
Biological: GSK Biologicals' Polio Sabin™ — 3 oral doses
  Other Names: OPV
Biological: GSK Biologicals' Zilbrix™ Hib — 3 IM doses.
  Other Names: DTPw-HBV/Hib vaccine

SUMMARY:
The purpose of this study is to assess the immunogenicity in terms of antibody response and the safety/reactogenicity in terms of solicited and unsolicited symptoms and serious adverse events following primary vaccination of African Sub-Saharan infants with pneumococcal conjugate vaccine GSK 1024850A co-administered with a diphtheria, tetanus, whole cell pertussis (DTPw)-combined vaccine and oral polio vaccine in children during the first 4 months of life.

DETAILED DESCRIPTION:
Vaccination course at 6, 10, 14 weeks of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including 6-10 weeks of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol should be enrolled in the study.
* Written or oral, signed or thumb-printed informed consent obtained from the parent(s)/guardian(s) of the child/ward. Where parent(s)/guardian(s) are illiterate, the consent form will be countersigned by a witness.
* Free of any known or suspected health problems (as established by medical history and clinical examination before entering into the study), that would contraindicate the initiation of routine immunizations outside a clinical trial context.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of the study vaccines, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* A family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period (Hepatitis B immunoglobulins at birth are allowed).
* Previous vaccination against, diphtheria, tetanus, pertussis, Haemophilus influenzae type b and/or Streptococcus pneumoniae.
* History of, or intercurrent diphtheria, tetanus, pertussis, hepatitis B, Streptococcus and Haemophilus influenzae type b disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment. Study entry should be delayed until the illness has improved.
* Babies for which birth weight is < 2 kilogram (if known) at Visit 1

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 365 (Actual)
Dates: Start 2008-06-18 (Actual); Primary Completion 2009-11-09 (Actual); Study Completion 2009-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Bamako, Mali
- GSK Investigational Site, Ikeja / Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=258

REFERENCES:
- [Background] Dicko A, Odusanya OO, Diallo AI, Santara G, Barry A, Dolo A, Diallo A, Kuyinu YA, Kehinde OA, Francois N, Borys D, Yarzabal JP, Moreira M, Schuerman L. Primary vaccination with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in infants in Mali and Nigeria: a randomized controlled trial. BMC Public Health. 2011 Nov 23;11:882. doi: 10.1186/1471-2458-11-882. PMID 22112189
- [Background] Odusanya OO, Kuyinu YA, Kehinde OA, Francois N, Yarzabal JP, Moreira M, Borys D, Schuerman L. Immunogenicity, safety and reactogenicity of the 10-valent pneumococcal non-typeable haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Nigerian Infants: a randomised trial. Niger Postgrad Med J. 2013 Dec;20(4):272-81. PMID 24633268
- [Background] Silfverdal SA, Coremans V, Francois N, Borys D, Cleerbout J. Safety profile of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Expert Rev Vaccines. 2017 Feb;16(2):109-121. doi: 10.1586/14760584.2016.1164044. Epub 2016 Sep 30. PMID 26954689
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At screening, the following steps occurred: check for inclusion/exclusion criteria, contraindications/ precautions, medical and vaccination history of the subjects and signing or thumb-printing informed consent forms.
Pre-assignment Details: Among 365 enrolled participants, 8 were not administered any study vaccine and hence were not considered as starting the study.
Period: Overall Study
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Started | 239 | 118
Completed | 231 | 116
Not Completed | 8 | 2
Not completed — Non-compliance with study procedures | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™ | Total
Number analyzed (Participants) | 239 | 118 | 357
Age, Continuous [Geometric Mean (Standard Deviation); unit: Weeks] | 7.1 (1.15) | 7 (1.18) | 7.07 (1.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 62 | 181
  Male | 120 | 56 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 239 | 118 | 357

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes
Description: Pneumococcal serotypes assessed were vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Seropositivity cut-off for the assay was an anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) concentrations greater than or equal to (≥) 0.05 microgram per milliliter (μg/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: The According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects with available immunogenicity data. The ATP cohort for immunogenicity included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 217 | 112
μg/mL
  Anti-1: number analyzed (Participants) | 217 | 108
  Anti-1 | 2.69 [2.42 to 2.99] | 0.03 [0.03 to 0.03]
  Anti-4 | 3.44 [3.06 to 3.87] | 0.03 [0.03 to 0.03]
  Anti-5: number analyzed (Participants) | 217 | 109
  Anti-5 | 4.17 [3.75 to 4.63] | 0.03 [0.03 to 0.04]
  Anti-6B | 0.95 [0.76 to 1.2] | 0.03 [0.03 to 0.03]
  Anti-7F: number analyzed (Participants) | 217 | 110
  Anti-7F | 3.33 [2.99 to 3.71] | 0.03 [0.03 to 0.04]
  Anti-9V | 2.39 [2.06 to 2.76] | 0.04 [0.03 to 0.05]
  Anti-14 | 3.8 [3.24 to 4.46] | 0.14 [0.11 to 0.17]
  Anti-18C | 10.01 [8.49 to 11.8] | 0.03 [0.03 to 0.04]
  Anti-19F: number analyzed (Participants) | 217 | 111
  Anti-19F | 7.65 [6.55 to 8.93] | 0.08 [0.07 to 0.1]
  Anti-23F | 1.1 [0.91 to 1.33] | 0.03 [0.03 to 0.04]

2. Primary Outcome: Antibody Concentrations Against Protein D (Anti-PD Antibodies)
Description: Anti-PD antibody concentrations were expressed in enzyme-linked immunsorbent assay (ELISA) units per milliliter (EL.U/mL). Seropositivity cut-off for the assay was an anti-PD antibody concentrations ≥ 100 EL.U/mL.
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 217 | 112
EL.U/mL | 3791.8 [3448.4 to 4169.3] | 85.4 [71.8 to 101.5]

3. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Anti-6A and -19A)
Description: Seropositivity status was defined as anti-pneumococcal cross-reactive serotypes 6A/19A antibody concentrations (Anti-6A/19A) ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 217 | 108
μg/mL
  Anti-6A | 0.09 [0.08 to 0.11] | 0.04 [0.04 to 0.05]
  Anti-19A | 0.15 [0.13 to 0.18] | 0.06 [0.05 to 0.07]

4. Secondary Outcome: Titers for Opsonophagocytic Activity (OPA) Against Vaccine Pneumococcal Serotypes
Description: Pneumococcal serotypes assessed were vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Seropositivity status was defined as an opsonophagocytic activity against vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (OPA-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) ≥ 8.
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 105 | 56
Titers
  OPA-1 | 83 [61.7 to 111.7] | 5 [3.8 to 6.4]
  OPA-4: number analyzed (Participants) | 105 | 55
  OPA-4 | 892.5 [759.4 to 1049] | 4.6 [3.9 to 5.5]
  OPA-5 | 82.7 [65.4 to 104.4] | 4.5 [3.8 to 5.2]
  OPA-6B: number analyzed (Participants) | 103 | 54
  OPA-6B | 538.6 [346 to 838.3] | 5.7 [4.1 to 7.9]
  OPA-7F: number analyzed (Participants) | 105 | 49
  OPA-7F | 2733 [2188.3 to 3413.3] | 31.5 [15.5 to 64]
  OPA-9V: number analyzed (Participants) | 105 | 54
  OPA-9V | 1023.7 [784.8 to 1335.2] | 8.4 [5.8 to 12.4]
  OPA-14: number analyzed (Participants) | 104 | 53
  OPA-14 | 1079.2 [776 to 1500.9] | 8.9 [5.7 to 14.1]
  OPA-18C | 617.6 [495.3 to 770] | 4.4 [3.8 to 5.2]
  OPA-19F | 358.3 [269.9 to 475.5] | 4.6 [3.8 to 5.7]
  OPA-23F: number analyzed (Participants) | 104 | 53
  OPA-23F | 881.8 [615 to 1264.4] | 6.6 [4.2 to 10.3]

5. Secondary Outcome: Titers for Opsonophagocytic Activity (OPA) Against Cross-reactive Pneumococcal Serotypes
Description: Pneumococcal serotypes assessed were cross-reactive pneumococcal serotypes 6A and 19A. Seropositivity status was defined as an opsonophagocytic activity against cross-reactive pneumococcal serotypes 6A and 19A (OPA-6A and 19A) ≥ 8.
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 105 | 56
Titres
  OPA-6A: number analyzed (Participants) | 101 | 56
  OPA-6A | 14.1 [9.4 to 21.2] | 6.1 [4.4 to 8.7]
  OPA-19A | 11 [8.3 to 14.6] | 4.3 [4 to 4.6]

6. Secondary Outcome: Number of Subjects Seropositive for Antibodies Against Vaccine Pneumococcal Serotypes
Description: Pneumococcal serotypes assessed were vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Seropositivity cut-off for the assay was an anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) concentrations ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 217 | 112
Participants
  Anti-1: number analyzed (Participants) | 217 | 108
  Anti-1 | 217 | 14
  Anti-4 | 217 | 12
  Anti-5: number analyzed (Participants) | 217 | 109
  Anti-5 | 217 | 18
  Anti-6B | 196 | 15
  Anti-7F: number analyzed (Participants) | 217 | 110
  Anti-7F | 217 | 19
  Anti-9V | 213 | 31
  Anti-14 | 217 | 91
  Anti-18C | 216 | 23
  Anti-19F: number analyzed (Participants) | 217 | 111
  Anti-19F | 217 | 73
  Anti-23F | 207 | 23

7. Secondary Outcome: Number of Subjects Seroprotected Against Vaccine Pneumococcal Serotypes
Description: Pneumococcal serotypes assessed were vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Seroprotection cut-off for the assay was an anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) concentrations ≥ 0.2 microgram per milliliter (μg/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 217 | 112
Participants
  Anti-1: number analyzed (Participants) | 217 | 108
  Anti-1 | 217 | 2
  Anti-4 | 217 | 3
  Anti-5: number analyzed (Participants) | 217 | 109
  Anti-5 | 217 | 4
  Anti-6B | 178 | 2
  Anti-7F: number analyzed (Participants) | 217 | 110
  Anti-7F | 216 | 2
  Anti-9V | 211 | 11
  Anti-14 | 215 | 40
  Anti-18C | 216 | 4
  Anti-19F: number analyzed (Participants) | 217 | 111
  Anti-19F | 214 | 25
  Anti-23F | 190 | 3

8. Secondary Outcome: Number of Subjects Seropositive for Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Anti-6A and -19A)
Description: Serotypes assessed were cross-reactive pneumococcal serotypes 6A and 19A. Seropositivity status was defined as anti-pneumococcal cross-reactive serotypes 6A/19A antibody concentrations (Anti-6A/19A) ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 217 | 108
Participants
  Anti-6A | 152 | 36
  Anti-19A | 176 | 49

9. Secondary Outcome: Number of Subjects Seroprotected Against Cross-reactive Pneumococcal Serotypes 6A and 19A (Anti-6A and -19A)
Description: Serotypes assessed were cross-reactive pneumococcal serotypes 6A and 19 A. Seroprotection cut-off for the assay was an anti-6A/19A antibody concentrations ≥ 0.2 microgram per milliliter (μg/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 217 | 108
Participants
  Anti-6A | 56 | 8
  Anti-19A | 95 | 15

10. Secondary Outcome: Number of Subjects Seropositive for Antibodies Against Protein D (Anti-PD Antibodies)
Description: Seropositivity cut-off for the assay was an anti-PD antibody concentrations ≥ 100 EL.U/mL.
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 217 | 112
Participants | 217 | 34

11. Secondary Outcome: Number of Subjects Seropositive for Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes
Description: as for outcome 4
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 105 | 56
Participants
  OPA-1 | 92 | 3
  OPA-4: number analyzed (Participants) | 105 | 55
  OPA-4 | 105 | 3
  OPA-5 | 100 | 2
  OPA-6B: number analyzed (Participants) | 103 | 54
  OPA-6B | 88 | 5
  OPA-7F: number analyzed (Participants) | 105 | 49
  OPA-7F | 105 | 21
  OPA-9V: number analyzed (Participants) | 105 | 54
  OPA-9V | 103 | 13
  OPA-14: number analyzed (Participants) | 104 | 53
  OPA-14 | 100 | 13
  OPA-18C | 103 | 2
  OPA-19F | 101 | 2
  OPA-23F: number analyzed (Participants) | 104 | 53
  OPA-23F | 97 | 5

12. Secondary Outcome: Number of Subjects Seropositive for Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes
Description: as for outcome 5
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 105 | 56
Participants
  OPA-6A: number analyzed (Participants) | 101 | 56
  OPA-6A | 31 | 6
  OPA-19A | 39 | 3

13. Secondary Outcome: Anti-Bordetella Pertussis (Anti-BPT) Antibody Concentrations
Description: Anti-BPT antibody concentrations were expressed in enzyme-linked immunosorbent assay (ELISA) unit per millilitre (EL.U/mL). Seropositivity cut-off for the assay was defined as an anti-BPT antibody concentrations ≥ 15 EL.U/mL
Time Frame: At Month 3, one month after the administration of the third dose of Synflorix vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 110 | 111
EL.U/mL | 111.9 [102 to 122.7] | 124.9 [111.7 to 139.7]

14. Secondary Outcome: Number of Subjects Seropositive for Antibodies Against Bordetella Pertussis (Anti-BPT)
Description: Seropositivity cut-off for the assay was defined as an anti-BPT antibody concentration ≥ 15 enzyme-linked immunosorbent assay (ELISA) unit per milliliter (EL.U/mL).
Time Frame: At Month 3, one month after the administration of the third dose of DTPw-HBV/Hib vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 110 | 111
Participants | 110 | 111

15. Secondary Outcome: Anti-diphtheria (Anti-D) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations
Description: The seroprotection cut-off for the assay was an anti-diphtheria toxoid or anti-tetanus toxoid antibody concentrations ≥ 0.1 international unit per milliliter (IU/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Tritanrix -HepB/ Hiberix vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 110 | 112
IU/mL
  Anti-D | 4.103 [3.527 to 4.773] | 3.13 [2.731 to 3.588]
  Anti-T | 6.484 [5.511 to 7.628] | 4.588 [3.88 to 5.426]

16. Secondary Outcome: Number of Subjects Seroprotected Against Diphtheria (D) and Tetanus Toxoids (TT) Antigens
Description: A subject seroprotected against D/TT antigens was defined as a subject with an Anti-D/-TT antibody concentration ≥ 0.1 IU/mL.
Time Frame: At Month 3, one month after the administration of the third dose of Tritanrix -HepB/ Hiberix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 110 | 112
Participants
  Anti-D | 110 | 112
  Anti-T | 110 | 112

17. Secondary Outcome: Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibody Concentrations
Description: Anti-PRP antibody concentrations were measured and tabulated in microgram per milliliter (μg/mL). Cut-off for the assay was ≥ 0.15 μg/mL.
Time Frame: At Month 3, one month after the administration of the third dose of Tritanrix -HepB/ Hiberix vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 110 | 112
μg/mL | 18.461 [14.256 to 23.907] | 10.137 [7.515 to 13.673]

18. Secondary Outcome: Number of Subjects Seroprotected Against Polyribosyl-ribitol Phosphate (PRP)
Description: Anti-PRP antibody concentrations were expressed in microgram per milliliter (μg/mL). The seroprotection cut-off applied for the assay was ≥ 0.15 μg/mL.
Time Frame: At Month 3, one month after the administration of the third dose of Tritanrix -HepB/ Hiberix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 110 | 112
Participants | 110 | 111

19. Secondary Outcome: Number of Subjects Seroprotected Against Polyribosyl-ribitol Phosphate (PRP) Antigens
Description: Anti-PRP antibody concentrations were expressed in microgram per milliliter (μg/mL). The seroprotection cut-off applied for the assay was ≥ 1 μg/mL.
Time Frame: At Month 3, one month after the administration of the third dose of Tritanrix -HepB/ Hiberix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 110 | 112
Participants | 107 | 102

20. Secondary Outcome: Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations
Description: The seroprotection cut-off for the endpoint was an anti-HBs antibody concentration ≥ 10 milli-international units per milliliter (mIU/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Tritanrix -HepB /Hiberix vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 91 | 96
mIU/mL | 1835.1 [1384 to 2433.2] | 1485.5 [1198.7 to 1840.9]

21. Secondary Outcome: Number of Subjects Seroprotected Against Anti-Hepatitis B Surface Antigens (HBs).
Description: The seroprotection cut-off values considered for this endpoint were an anti-HBs antibody concentration ≥ 10 and 100 milli-international units per milliliter (mIU/mL).
Time Frame: At Month 3, one month after the administration of the third dose of Tritanrix HepB/ Hiberix vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 91 | 96
Participants
  Anti-HBs ≥ 10 mIU/mL | 89 | 96
  Anti-HBs ≥ 100 mIU/mL | 89 | 94

22. Secondary Outcome: Number of Subjects With Any and Any Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed included pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/ spontaneously painful. Grade 3 swelling/ redness was defined as swelling/ redness greater than (>) 30 millimeters (mm). "Any" was defined as incidence of the specified symptom regardless of intensity.
Time Frame: Within the 4-day (Days 0 to 3) follow-up periods after each vaccination, across doses and across vaccines
Population: The Total Vaccinated Cohort included all evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 239 | 118
Participants
  Any Pain | 234 | 112
  Grade 3 Pain | 8 | 3
  Any Redness | 57 | 30
  Grade 3 Redness | 0 | 0
  Any Swelling | 173 | 83
  Grade 3 Swelling | 22 | 11

23. Secondary Outcome: Number of Subjects With Any and Any Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever (defined as rectal temperature ≥ 38.0°C), irritability, and loss of appetite. "Any" was defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (rectal temperature) greater than (>) 40.0 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/ preventing normal activity. Grade 3 loss of appetite was defined as the subject not eating at all.
Time Frame: Within the 4-day (Days 0 to 3) follow-up periods after each vaccination, across doses and across vaccines
Population: The Total Vaccinated Cohort included all evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 239 | 118
Participants
  Any Drowsiness | 24 | 12
  Grade 3 Drowsiness | 0 | 0
  Any Fever (Rectally) | 207 | 105
  Grade 3 Fever (Rectally) | 1 | 0
  Any Irritability | 192 | 88
  Grade 3 Irritability | 6 | 2
  Any Loss of appetite | 37 | 15
  Grade 3 Loss of appetite | 1 | 0

24. Secondary Outcome: Number of Subjects With Fever (Temperature Measured Rectally) > the Cut-off
Description: The cut-off for the assay was > 39.0°C.
Time Frame: Within the 4-day (Days 0 to 3) follow-up periods after each vaccination, across doses and across vaccines
Population: The Total Vaccinated Cohort included all evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 239 | 118
Participants | 40 | 13

25. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" was defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) follow-up periods post vaccination, across doses and across vaccines
Population: The Total Vaccinated Cohort included all evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 239 | 118
Participants | 176 | 92

26. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/ incapacity.
Time Frame: Throughout the entire study period, from Month 0 to Month 3
Population: The Total Vaccinated Cohort included all evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
Number analyzed (Participants) | 239 | 118
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms and unsolicited AEs: During the 4-day (Days 0-3) and 31-day (Days 0-30) post vaccination follow-up periods, respectively, across doses and across vaccines. SAEs: throughout the entire study period, from Month 0 to Month 3
Arm/Group | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ | Zilbrix™ Hib + Polio Sabin™
All-Cause Mortality (participants affected / at risk) | 0/239 | 0/118
Serious Adverse Events (participants affected / at risk) | 5/239 | 0/118
Other Adverse Events (participants affected / at risk) | 238/239 | 117/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ (N=239) | Zilbrix™ Hib + Polio Sabin™ (N=118)
Bronchopneumonia (Vascular disorders) | 4 | 0
Haematoma (Vascular disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix™ + Zilbrix™ Hib + Polio Sabin™ (N=239) | Zilbrix™ Hib + Polio Sabin™ (N=118)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 83 | 46
Conjunctivitis (Eye disorders) | 35 | 16
Pain (General disorders) | 234 | 112
Redness (General disorders) | 57 | 30
Swelling (General disorders) | 173 | 83
Drowsiness (General disorders) | 24 | 12
Fever (rectal temperature ≥ 38.5°C) (General disorders) | 207 | 105
Irritability (General disorders) | 192 | 88
Loss of appetite (General disorders) | 37 | 15
Injection site erosion (General disorders) | 1 | 6
Injection site induration (General disorders) | 22 | 20
Abdominal distension (Gastrointestinal disorders) | 43 | 22
Gastrointestinal disorder (Gastrointestinal disorders) | 25 | 15
Stomatitis (Gastrointestinal disorders) | 13 | 4
Bronchitis (Infections and infestations) | 12 | 6
Ear infection (Infections and infestations) | 42 | 21
Gastroenteritis (Infections and infestations) | 61 | 32
Pharyngitis (Infections and infestations) | 14 | 5
Respiratory tract infection (Infections and infestations) | 17 | 11
Rhinitis (Infections and infestations) | 85 | 42
Skin infection (Infections and infestations) | 16 | 16
Urinary tract infection (Infections and infestations) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.